CLINICAL TRIAL: NCT03996590
Title: WATCH (Wessex AsThma CoHort of Difficult Asthma): A Longitudinal Cohort Study to Facilitate Better Understanding and Management of Difficult Asthma Encountered in Clinical Practice
Brief Title: Wessex Asthma Cohort of Difficult Asthma
Acronym: WATCH
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Novartis (Industry); Boehringer Ingelheim (Industry); National Institutes of Health (NIH) (NIH); Owlstone Ltd (Industry); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: RHM MED1216
Record Dates: First submitted 2019-06-20; First posted 2019-06-25 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Asthma
Keywords: Difficult Asthma; Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 35 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asthma is now widely recognised to be a heterogeneous disease. The last two decades have seen the identification of a number of biological targets and development of various novel therapies. Despite this, asthma still represents a significant health and economic burden worldwide. Why some individuals should continue to suffer remains unclear.

The Wessex Asthma Cohort of Difficult Asthma (WATCH) is an ongoing 'real-life', prospective study of patients in the University Hospital Southampton Foundation Trust (UHSFT) Difficult Asthma service. Research data capture is aligned with the extensive clinical characterisation required of a commissioned National Health Service (NHS) Specialist Centre for Severe Asthma. Data acquisition includes detailed clinical, health and disease-related questionnaires, anthropometry, allergy and lung function testing, radiological imaging (in a small subset) and collection of biological samples (blood, urine and sputum). Prospective data are captured in parallel to clinical follow up appointments, with data entered into a bespoke database.

The pragmatic ongoing nature of the WATCH study allows comprehensive assessment of the real world clinical spectrum seen in a Specialist Asthma Centre and allows a longitudinal perspective of deeply phenotyped patients. It is anticipated that the WATCH cohort would act as a vehicle for potential collaborative asthma studies and will build upon our understanding of mechanisms underlying difficult asthma.

DETAILED DESCRIPTION:
Asthma is estimated to affect 5.2 million people in the United Kingdom (UK), half of whom experience severe symptoms at some point in their lives, and 500,000 of whom may be unresponsive to currently available therapies (Asthma UK; "living on a knife edge" 2004). Severe Asthma probably accounts for 80% of asthma-related health expenditure (Chung KF, Eur Res Mon 2003, 23: 313). In this regard it is estimated to directly cost the NHS (National Health Service) £1 billion per year but also poses considerable hidden societal costs through disability, missed schooling and lost work days.

While Severe Asthma is a significant health-economic problem, the availability of effective treatments in clinical practice remains limited. However there is a growing realisation of the heterogeneity of asthma, which is not a single condition, but composed of numerous potential phenotypes (Wenzel S Nat Med 2012 18(5):716-25) some of which may show association to more severe disease status. In this regard recent adoption of unbiased statistical techniques such as cluster analysis has consistently demonstrated presence of severe asthma clusters in both adult and paediatric populations. These clinical phenotypes may show specific pathophysiological associations leading to classification of endotypes. Accompanying this growing understanding of the diverse nature of asthma is the realisation that there are also a diverse range of treatment responses dependent on the underlying nature of an individual's disease. This naturally leads to the concept of personalised therapy regimes for patients with Severe Asthma that better target their individual disease. Omalizumab is the first biological asthma treatment to meet that need in patients with severe allergic asthma. Numerous potential biological agents are in development that show promise in targeting patients with particular disease phenotypes/ endotypes such as mepolizumab, lebrikizumab and dupilimumab.

The organisation of Clinical Services for Severe Asthma is undergoing major change with the initiation of Specialised Commissioning of such Services by NHS England in 2014. A core requirement for Specialist Centres being Commissioned under this process will be the maintenance of accurate clinical disease registers which link to the BTS Difficult Asthma Registry and support collaborative research studies in the future.

The Difficult Asthma Clinics at Southampton and Portsmouth currently care for 1000 and 400 patients with problematic disease respectively. The two asthma services already collaborate as the Wessex Asthma Network to provide education across the Wessex region. Both services in their roles as Commissioned Specialist Clinical Centre for Severe Asthma receive regional referrals from a wide geographical area. We intend to initiate a comprehensively assessed Difficult Asthma Cohort by inviting all patients in our clinics to participate and contribute data gained through their clinical assessment. This would support ongoing contribution to research via the BTS Difficult Asthma Registry. In addition, a real-life clinical characterisation of Difficult Asthma would provide the basis for a better understanding of the nature of that disease relevant to clinical practice. It would also provide opportunity to develop a better endotype defined understanding of Difficult Asthma that facilitates stratified development of more effective treatment strategies. The Cohort will become a resource for future therapeutic studies in Difficult Asthma with Cohort participants being invited to consent separately into those studies based upon their characterisation through the Cohort.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the Adult or Transitional Regional Asthma Clinics at participating hospitals.
* On high-dose therapies, with or without the addition of continuous or frequent use of oral steroids (or steroid sparing therapies), as defined by the BTS (British Thoracic Society) Adult Asthma Management Guidelines (2016).

Exclusion Criteria:

* Asthma patients who are not referred to the Adult or Transitional Regional Asthma Clinics at participating hospitals.
* Any patients who are not on high-dose therapies, with or without the addition of continuous or frequent use of oral steroids (or steroid sparing therapies), as per the BTS (British Thoracic Society) Adult Asthma Management Guidelines (2016).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe or difficult asthma referred to secondary and tertiary referral centres
Sampling Method: Non-Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Cohort Characterisation | 35 years
  To develop a phenotypic characterisation of the heterogeneous nature of severe asthma seen in clinical practice that reflects disease natural history and treatment intervention responsiveness

SECONDARY OUTCOMES:
Clinical Endotyping | 35 years
  To relate well characterised clinical disease phenotypes to pathophysiological endotypes of severe asthma.
Patient Stratification | 35 years
  To enable accurate stratification of patients for trials of novel pharmacological and non-pharmacological treatment strategies that facilitates an era of individualised patient management.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh J Kurukulaaratchy, DM FRCP, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Portsmouth Hospitals NHS Trust, Portsmouth, Hamsphire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hamsphire
  - Isle of Wight NHS Trust, Newport, Isle Of Wight

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith DH, Malone DC, Lawson KA, Okamoto LJ, Battista C, Saunders WB. A national estimate of the economic costs of asthma. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):787-93. doi: 10.1164/ajrccm.156.3.9611072. PMID 9309994
- [Background] Barnes PJ, Jonsson B, Klim JB. The costs of asthma. Eur Respir J. 1996 Apr;9(4):636-42. doi: 10.1183/09031936.96.09040636. PMID 8726924
- [Background] Masoli M, Fabian D, Holt S, Beasley R; Global Initiative for Asthma (GINA) Program. The global burden of asthma: executive summary of the GINA Dissemination Committee report. Allergy. 2004 May;59(5):469-78. doi: 10.1111/j.1398-9995.2004.00526.x. No abstract available. PMID 15080825
- [Background] Wenzel SE. Asthma phenotypes: the evolution from clinical to molecular approaches. Nat Med. 2012 May 4;18(5):716-25. doi: 10.1038/nm.2678. PMID 22561835
- [Background] Moore WC, Meyers DA, Wenzel SE, Teague WG, Li H, Li X, D'Agostino R Jr, Castro M, Curran-Everett D, Fitzpatrick AM, Gaston B, Jarjour NN, Sorkness R, Calhoun WJ, Chung KF, Comhair SA, Dweik RA, Israel E, Peters SP, Busse WW, Erzurum SC, Bleecker ER; National Heart, Lung, and Blood Institute's Severe Asthma Research Program. Identification of asthma phenotypes using cluster analysis in the Severe Asthma Research Program. Am J Respir Crit Care Med. 2010 Feb 15;181(4):315-23. doi: 10.1164/rccm.200906-0896OC. Epub 2009 Nov 5. PMID 19892860
- [Background] Haldar P, Pavord ID, Shaw DE, Berry MA, Thomas M, Brightling CE, Wardlaw AJ, Green RH. Cluster analysis and clinical asthma phenotypes. Am J Respir Crit Care Med. 2008 Aug 1;178(3):218-224. doi: 10.1164/rccm.200711-1754OC. Epub 2008 May 14. PMID 18480428
- [Background] Weatherall M, Travers J, Shirtcliffe PM, Marsh SE, Williams MV, Nowitz MR, Aldington S, Beasley R. Distinct clinical phenotypes of airways disease defined by cluster analysis. Eur Respir J. 2009 Oct;34(4):812-8. doi: 10.1183/09031936.00174408. Epub 2009 Apr 8. PMID 19357143
- [Background] Fitzpatrick AM, Teague WG, Meyers DA, Peters SP, Li X, Li H, Wenzel SE, Aujla S, Castro M, Bacharier LB, Gaston BM, Bleecker ER, Moore WC; National Institutes of Health/National Heart, Lung, and Blood Institute Severe Asthma Research Program. Heterogeneity of severe asthma in childhood: confirmation by cluster analysis of children in the National Institutes of Health/National Heart, Lung, and Blood Institute Severe Asthma Research Program. J Allergy Clin Immunol. 2011 Feb;127(2):382-389.e1-13. doi: 10.1016/j.jaci.2010.11.015. Epub 2010 Dec 31. PMID 21195471
- [Background] Just J, Gouvis-Echraghi R, Rouve S, Wanin S, Moreau D, Annesi-Maesano I. Two novel, severe asthma phenotypes identified during childhood using a clustering approach. Eur Respir J. 2012 Jul;40(1):55-60. doi: 10.1183/09031936.00123411. Epub 2012 Jan 20. PMID 22267763
- [Background] Lotvall J, Akdis CA, Bacharier LB, Bjermer L, Casale TB, Custovic A, Lemanske RF Jr, Wardlaw AJ, Wenzel SE, Greenberger PA. Asthma endotypes: a new approach to classification of disease entities within the asthma syndrome. J Allergy Clin Immunol. 2011 Feb;127(2):355-60. doi: 10.1016/j.jaci.2010.11.037. PMID 21281866
- [Background] Pavord ID, Korn S, Howarth P, Bleecker ER, Buhl R, Keene ON, Ortega H, Chanez P. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):651-9. doi: 10.1016/S0140-6736(12)60988-X. PMID 22901886
- [Background] Corren J, Lemanske RF, Hanania NA, Korenblat PE, Parsey MV, Arron JR, Harris JM, Scheerens H, Wu LC, Su Z, Mosesova S, Eisner MD, Bohen SP, Matthews JG. Lebrikizumab treatment in adults with asthma. N Engl J Med. 2011 Sep 22;365(12):1088-98. doi: 10.1056/NEJMoa1106469. Epub 2011 Aug 3. PMID 21812663
- [Background] Wenzel S, Ford L, Pearlman D, Spector S, Sher L, Skobieranda F, Wang L, Kirkesseli S, Rocklin R, Bock B, Hamilton J, Ming JE, Radin A, Stahl N, Yancopoulos GD, Graham N, Pirozzi G. Dupilumab in persistent asthma with elevated eosinophil levels. N Engl J Med. 2013 Jun 27;368(26):2455-66. doi: 10.1056/NEJMoa1304048. Epub 2013 May 21. PMID 23688323
- [Derived] Mistry H, Ajsivinac Soberanis HM, Kyyaly MA, Azim A, Barber C, Knight D, Newell C, Haitchi HM, Wilkinson T, Howarth P, Seumois G, Vijayanand P, Arshad SH, Kurukulaaratchy RJ. The Clinical Implications of Aspergillus Fumigatus Sensitization in Difficult-To-Treat Asthma Patients. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4254-4267.e10. doi: 10.1016/j.jaip.2021.08.038. Epub 2021 Sep 14. PMID 34534722

DOCUMENTS (1):
  • Informed Consent Form (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT03996590/ICF_000.pdf